CLINICAL TRIAL: NCT00914550
Title: Use Of Procalcitonin Level For Guidance of The Treatment of Suspected Community Acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Michael S. Niederman, M.D., Principal Investigator, Winthrop University Hospital
Other Study IDs: 107003-3
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Pneumonia; Radiographic Lung Infiltrates
Keywords: Pneumonia; Lung Infiltrates; Antibiotic discontinuation; De-escalation therapy
MeSH Terms: conditions — Pneumonia | interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum Procalcitonin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Procalcitonin level, caregiver informed: Procalcitonin level for patients with lung infiltrates:caregivers know/ do not know results
  Interventions: Other: Procalcitonin level, caregiver informed

INTERVENTIONS:
Other: Procalcitonin level, caregiver informed — Procalcitonin levels will be measured and known by investigator, only 1/2 of the patients' caregivers will know the results of serial Procalcitonin levels. We will analyze the rate of antibiotic discontinuation for the two arms

SUMMARY:
The purpose of the study is to learn if a blood test is helpful to the doctors in deciding whether you need antibiotic therapy for possible pneumonia. The blood test is called a Procalcitonin level and sometimes the test reflects infection with certain bacteria (germs). When the doctors learn the results of these blood tests, they may be able to stop some of the antibiotic medications that they may have given to the patients. The study is designed, so that on a randomized basis (50/50 chance) the results from measuring Procalcitonin will be given to the patients' doctor. When the doctor receives these results, he/she may use this information, along with other information, to decide whether to continue antibiotic therapy.

DETAILED DESCRIPTION:
To evaluate the usefulness of serum Procalcitonin level measured to guide the antibiotic treatment of patients with radiographic lung infiltrates.The subjects involved in the study will be divided in two arms ,study arm where the caregivers will know the result of Procalcitonin level and they can change /withheld the antibiotic for the subjects.In other arm only investigators will know the Procalcitonin level. We expect to enroll 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* New radiographic findings consistent with the presence of infiltrates
* Antibiotic therapy

Exclusion Criteria:

* Critically ill patients on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to Winthrop University Hospital with Lung Infiltrates undergoing antibiotic therapy
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Differences in antibiotic discontinuation as an effect of the caregivers learning Procalcitonin levels for the therapy of new radiographic lung infiltrates | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Niederman, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Niederman MS. Making sense of scoring systems in community acquired pneumonia. Respirology. 2009 Apr;14(3):327-35. doi: 10.1111/j.1440-1843.2009.01494.x. PMID 19353770
- [Background] Menendez R, Martinez R, Reyes S, Mensa J, Filella X, Marcos MA, Martinez A, Esquinas C, Ramirez P, Torres A. Biomarkers improve mortality prediction by prognostic scales in community-acquired pneumonia. Thorax. 2009 Jul;64(7):587-91. doi: 10.1136/thx.2008.105312. Epub 2009 Jan 8. PMID 19131448
- [Background] Niederman MS. Biological markers to determine eligibility in trials for community-acquired pneumonia: a focus on procalcitonin. Clin Infect Dis. 2008 Dec 1;47 Suppl 3:S127-32. doi: 10.1086/591393. PMID 18986278
- [Background] Haeuptle J, Zaborsky R, Fiumefreddo R, Trampuz A, Steffen I, Frei R, Christ-Crain M, Muller B, Schuetz P. Prognostic value of procalcitonin in Legionella pneumonia. Eur J Clin Microbiol Infect Dis. 2009 Jan;28(1):55-60. doi: 10.1007/s10096-008-0592-5. Epub 2008 Aug 2. PMID 18677519
- [Background] Menendez R, Cavalcanti M, Reyes S, Mensa J, Martinez R, Marcos MA, Filella X, Niederman M, Torres A. Markers of treatment failure in hospitalised community acquired pneumonia. Thorax. 2008 May;63(5):447-52. doi: 10.1136/thx.2007.086785. Epub 2008 Feb 1. PMID 18245147
- [Background] Ramirez P, Garcia MA, Ferrer M, Aznar J, Valencia M, Sahuquillo JM, Menendez R, Asenjo MA, Torres A. Sequential measurements of procalcitonin levels in diagnosing ventilator-associated pneumonia. Eur Respir J. 2008 Feb;31(2):356-62. doi: 10.1183/09031936.00086707. Epub 2007 Oct 24. PMID 17959634
- [Background] Schuetz P, Christ-Crain M, Wolbers M, Schild U, Thomann R, Falconnier C, Widmer I, Neidert S, Blum CA, Schonenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Muller B; ProHOSP study group. Procalcitonin guided antibiotic therapy and hospitalization in patients with lower respiratory tract infections: a prospective, multicenter, randomized controlled trial. BMC Health Serv Res. 2007 Jul 5;7:102. doi: 10.1186/1472-6963-7-102. PMID 17615073
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- See also: Guidelines on the management of Community-acquired Pneumonia by Infections Diseases Society of America and American Thoracic Society — http://thoracic.org/statements/resources/mtpi/idsaats-cap.pdf